CLINICAL TRIAL: NCT06084299
Title: Immunotherapy Using Tumor Infiltrating Lymphocytes for Patients With Advanced Liver Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhiyong Huang (Other)
Collaborators: Wuhan Elongevity Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Zhiyong Huang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YS-TIL-TJL01
Record Dates: First submitted 2023-10-03; First posted 2023-10-16 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (autologous tumor infiltrating lymphocytes) (Experimental): Post-NMA lymphodepletion, patients are infused with their autologous TIL followed by IL-2 administration.
  Interventions: Biological: Autologous Tumor Infiltrating Lymphocytes

INTERVENTIONS:
Biological: Autologous Tumor Infiltrating Lymphocytes — Fresh tumor samples will be resected from enrolled patients. Autologous TILs will be extracted and reinfused to corresponding patients after ex vivo stimulation, activation, and extensive expansion.

SUMMARY:
Single-arm, open-label, interventional study evaluating adoptive cell therapy (ACT) with autologous tumor-infiltrating lymphocytes (TIL) infusion followed by IL-2 after a non-myeloablative(NMA) lymphodepletion preparative regimen for the treatment of patients with advanced liver cancer.

DETAILED DESCRIPTION:
This is an adoptive cell transfer therapy that utilizes an autologous TIL manufacturing process for the treatment of patients with advanced liver cancer. The cell transfer therapy used in this study involves patients receiving a non-myeloablative lymphodepletion preparative regimen, followed by i.v. infusion of autologous tumor-infiltrating lymphocytes followed by the administration of a regimen of IL-2.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must be informed of the study before the test and voluntarily sign a written informed consent.
* Age of the patients was between 18~70 years
* Eligible patients have histologically proven advanced liver cancer
* Eastern Cooperative Oncology Group (ECOG) performance status was 0-1
* Metastatic lesions are confirmed by PET-CT, CT, MR and/or intraoperative exploration (more than 3, at least one accessible metastasis to procure for TILs)
* Patients have at least one separate additional measurable tumour lesion according to RECIST version 1.1 standard.
* The disease has progressed after at least two previous lines of standard treatment and there is no effective treatment option available
* Adequate normal organ and marrow function were present, including absolute neutrophil count ≥ 1×10^9/L, leukocyte count ≥ 3×10^9/L, platelet count ≥ 75×10^9/L, hemoglobin ≥ 80 g/L, AST and ALT ≤ 2× of upper limit of normal, Serum creatinine ≤ 1.5× upper normal limits, Serum total bilirubin ≤ 1.5× upper normal limits
* Female subjects of childbearing age must have a negative urine or serum HCG test within 7 days before cell reinfusion
* Provide at least one gram of fresh tumor tissue and 10ml of peripheral blood for whole exome sequencing and TIL isolation and culture.
* Expected survival was at least 3 months
* Child-Push liver function score grade is A within seven days before the cell reinfusion.

Exclusion Criteria:

* With previous or concurrent other active cancer (except carcinoma in situ that has been cured without onset within 5 years, or those that can be cured by adequate treatment)
* Patients with metastasis to Central Nervous System or brain
* Have received organ transplantation in the past
* Received major liver surgery within 4 weeks before the first administration (except liver metastases biopsy).
* Received local treatment of the liver or other parts within 4 weeks before the first administration (transcatheter arterial chemoembolization [TACE], transcatheter arterial embolization [TAE], hepatic artery infusion [HAI], radiotherapy, radioembolization or ablation). Subjects are not eligible to participate in the study if the above-mentioned treatment is carried out between the last dose of sorafenib or oxaliplatin-containing regimen and the first study administration.
* After CT angiography examination, there is severe arterial embolism or hepatic artery vascular variation.
* APTT or PT >= 5 UNL, or with bleeding evidence in two months or bleeding history in prior to the clinical study, no matter how serious it is
* Active inflammation within 7 days after systemic antibiotics treatment
* Subjects who have undergone major surgery or severe trauma such as laparotomy, thoracotomy, and laparoscopic organ removal within 4 weeks before enrollment.
* Active coronary artery disease, serious or unstable angina pectoris, or newly diagnosed angina pectoris or myocardial infarction within 12 months prior to the clinical study
* Thrombosis or embolism event within 12 months prior to the clinical study, such as cerebrovascular accident ( including TIA) or pulmonary embolism
* Congestive heart failure of NYHA >= Class II
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml C Hepatitis, defined as HCV-RNA higher than the detection limit of the analytical method) or co-infection with hepatitis B and hepatitis C.
* Presence of any active, known or suspected autoimmune disease. Subjects in a stable state who do not require systemic immunosuppressive therapy are allowed, such as: type 1 diabetes mellitus, hypothyroidism requiring only hormone replacement therapy, and skin diseases that do not require systemic therapy (e.g., vitiligo, psoriasis disease and hair loss).
* Any interstitial lung disease, noninfectious causes of lung inflammation, or uncontrolled systemic disease (e.g. diabetes, pulmonary fibrosis, or acute pneumonia)
* Any adverse event of CTCAE (Ver 5.0) grade 2 or higher induced by previous treatment, except anemia, hair loss, and skin pigmentation
* Pregnant or lactating women or those who are positive in pregnancy test before 1st injection
* The investigator believes that the subject has any clinical or laboratory abnormalities or compliance problems and is not suitable for participating in this clinical study.
* With serious psychological or mental abnormalities
* Joined other clinical trials in four weeks prior to this study
* Patients who have a history of hypersensitivity to cyclophosphamide and fludarabine.
* Other researchers think that they are not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Types and incidence of Dose-limiting toxicity (DLT) [Safety and Tolerability] | 1 month
  Dose-limiting toxicity (DLT) will be collected and graded according to CTCAE v5.0
Types and incidence of adverse events (AEs) ,serious adverse events (SAEs) [Safety and Tolerability] | Up to 24 months
  AE will be collected and graded according to CTCAE v5.0
Maximum tolerated dose [Safety and Tolerability] | 1 month
  Evaluate the maximum tolerated dose of TILs in patients with advanced liver cancer

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 6 months
  PFS will be calculated as the time from TIL infusion to disease progression or death from any cause (whichever occurs first) (RECIST v1.1).
Disease Control Rate (DCR) | Up to 24 months
  DCR will be calculated as the percentage of patients who achieved Stable Disease(SD) or better for more than 8 weeks (RECIST v1.1).
Objective response rate (ORR) | Up to 24 months
  ORR will be calculated as the percentage of patients who achieved partial response (PR) or better (RECIST v1.1).
Overall Survival (OS) | Up to 24 months
  Time from TIL infusion to time of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Huang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chesney J, Lewis KD, Kluger H, Hamid O, Whitman E, Thomas S, Wermke M, Cusnir M, Domingo-Musibay E, Phan GQ, Kirkwood JM, Hassel JC, Orloff M, Larkin J, Weber J, Furness AJS, Khushalani NI, Medina T, Egger ME, Graf Finckenstein F, Jagasia M, Hari P, Sulur G, Shi W, Wu X, Sarnaik A. Efficacy and safety of lifileucel, a one-time autologous tumor-infiltrating lymphocyte (TIL) cell therapy, in patients with advanced melanoma after progression on immune checkpoint inhibitors and targeted therapies: pooled analysis of consecutive cohorts of the C-144-01 study. J Immunother Cancer. 2022 Dec;10(12):e005755. doi: 10.1136/jitc-2022-005755. PMID 36600653